CLINICAL TRIAL: NCT04126863
Title: Omphaloceles and Associated Malformations in Preterm and Term Newborns
Brief Title: Omphaloceles and Associated Malformations
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: 425/2019BO1
Record Dates: First submitted 2019-09-19; First posted 2019-10-15 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2022-05

CONDITIONS: Omphalocele
MeSH Terms: conditions — Hernia, Umbilical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Major birth defects like omphalocele are diagnosed in 3-8% of all newborns in Germany each year. Prevention and treatment quality of congenital malformations are key concerns for child health. Poor long-term outcome is more likely in the presence of associated structural or chromosomal abnormalities that occur in approximately 50-77% of these infants. Furthermore, many newborns have respiratory failure and supposedly pulmonary hypertension - another reason for increased mortality.

As part of the Surveillance Unit for Rare Pediatric Conditions in Germany (Erhebungseinheit für seltene pädiatrische Erkrankungen in Deutschland), all neonatological departments receive over two years monthly reporting cards to notify the study centre of cases, which will be analysed based on anonymised questionnaires.

DETAILED DESCRIPTION:
An observational study using anonymized questionnaires, enrolled over two years (01/07/2019 - 30/06/2021) via the Surveillance Unit for Rare Pediatric Conditions in Germany (ESPED - Erhebungseinheit für seltene pädiatrische Erkrankungen in Deutschland). The nationwide epidemiological data collection contents information about the incidence of omphalocele, associated malformations and risk factors for the occurrence of omphalocele, especially for pulmonary hypertension and its treatment.

We use the following inclusion criteria: preterm and term babies' ≤ 28 days of life.

The aim of our study is a reliable, population-related data acquisition about prevalence of omphalocele, associated malformations and possible risk factors and characteristic early warning symptoms regarding concomitant diseases. Thereby, in the future it will be possible to develop prevention strategies für early detection and treatment of omphalocele and the associated malformations/ diseases to improve outcome for these babies. A further aim is to follow-up the thriving and the psychomotor development of these babies in the age of two years.

ELIGIBILITY:
Inclusion Criteria:

* preterm and term newborns ≤ 28 days
* present omphalocele

Exclusion Criteria:

* none

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm and term babies with omphalocele ≤ 28 days of life
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with Omphalocele | two years
  Collection of data to calculate the prevalence of omphaloceles
Number of patients with omphaloceles and associated malformations, especially pulmonary hypertension | two years
  Collection of data to calculate the prevalence of omphalocele associated malformations
Two-years outcome | two years
  Monitoring of weighting and thriving and of psychomotor development on the basis of a general developmental screening tool (ages & stages questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Poets, Prof., Study Director — University Childrens Hospital Tübingen
Locations (1):
- Department of Neonatology, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No